CLINICAL TRIAL: NCT05412576
Title: a Pilot Randomized Controlled Trial on the Safety and Efficacy of Different Doses of Lidocaine Infusion for Postoperative Analgesia in Elderly Patients With Colorectal Cancer Surgery
Brief Title: a Pilot Study of Lidocaine Infusion for Postoperative Analgesia in Elderly Patients With Colorectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-1180
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IVL0.5 group (Experimental): At the beginning of surgery, lidocaine 0.5mg/kg per hour will be continuously infused (using ideal body weight) and stopped at the end of the procedure.
  Interventions: Drug: Lidocaine Hydrochloride 2% Injection Solution
- IVL1.0 group (Experimental): At the beginning of surgery, lidocaine 0.5mg/kg per hour will be continuously infused (using ideal body weight) and stopped at the end of the procedure.
  Interventions: Drug: Lidocaine Hydrochloride 2% Injection Solution
- IVL1.5 group (Experimental): At the beginning of surgery, lidocaine 0.5mg/kg per hour will be continuously infused (using ideal body weight) and stopped at the end of the procedure.
  Interventions: Drug: Lidocaine Hydrochloride 2% Injection Solution
- Placebo group (Placebo Comparator): At the beginning of surgery, in the placebo group, the same dose of normal saline as the experimental groups will be given until the procedure is over.
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: Lidocaine Hydrochloride 2% Injection Solution — Injectable
  Other Names: IVL 0.5/1.0/1.5group
  Arms: IVL0.5 group; IVL1.0 group; IVL1.5 group
Drug: 0.9% NaCl — Injectable
  Other Names: placebo group
  Arms: Placebo group

SUMMARY:
patients who meet the enrollment criteria will be randomized 1:1:1:1 to the different doses of lidocaine or the placebo group. In the lidocaine groups, at the beginning of surgery, lidocaine 0.5mg/kg, 1.0mg/kg, and 1.5mg/kg per hour were continuously infused (using ideal body weight) respectively during the whole procedure. In contrast, the control group was infused with the same dose of normal saline. All the infusion procedures will be stopped at the end of surgery

DETAILED DESCRIPTION:
patients who meet the enrollment criteria will be randomized 1:1:1:1 to the different doses of lidocaine or the placebo group. In the lidocaine groups, at the beginning of surgery, lidocaine 0.5mg/kg, 1.0mg/kg, and 1.5mg/kg per hour were continuously infused (using ideal body weight) respectively during the whole procedure. In contrast, the control group was infused with the same dose of normal saline. All the infusion procedures will be stopped at the end of surgery. Subsequently, all subjects will receive an analgesic device named Patient-Controlled Intravenous Analgesia pump, briefly, PCIA pump during the first 72 postoperative hours. PCIA pump contains lidocaine 30mg/kg, sufentanil 2 μg/kg, and granisetron 12 mg diluted to 200 mL in 0.9 % normal saline, while in the placebo group, the lidocaine will be replaced with the equal dose of 0.9% normal saline and other components unchanged. All the background infusions of PCIA will be set at 2 ml/h, the bolus volume of each PCIA press is 2 ml and the lockout interval is 15 min.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years old；
* American Society Anesthesiologygist(ASA)I~III；
* Patients scheduled for colorectal cancer surgery；
* The surgery takes more than two hours

Exclusion Criteria:

* BMI≥30kg/㎡or BMI≤18kg/㎡；
* Combined with other organ malignancies；
* Chronic opioid use, substance abuse, contraindication to the use or incompatibility of any drug in the study；
* Patients with liver and kidney insufficiency and chronic pain at the surgical site；
* Accompanied by severe heart disease (such as severe atrioventricular block, severe heart failure, etc.)；
* A history of uncontrolled seizures or acute porphyria；
* Patients who have taken other experimental drugs or participated in or are participating in other clinical trials within 3 months before being enrolled in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
The incidence of moderate to severe pain (NRS score≥4）during movement (i.e.deep breathing) 24 hours after surgery | The first 24 hours after surgery
  The pain is evaluated using a numbering rating score(NRS).NRS scores range from 0 to 10 points, with 0 points repressing no pain,1-3points repressing mild pain, 4-6 points repressing moderate pain, 7-9 points repressing severe pain, and 10 points repressing the strongest pain.

SECONDARY OUTCOMES:
The blood concentration of lidocaine immediately and 24 hours after the operation | immediately after the operation; 24 hours after the operation
  Immediately after the operation and 24 hours after the procedure, the researchers drew 3ml of blood respectively from patients to detect the blood concentration of lidocaine.
The incidence of moderate to severe pain 24 hours after surgery at rest, 48 and 72 hours after surgery, both at rest and during movement | 24 hours after surgery at rest; 48 and 72 hours after surgery, both at rest and during movement
  The pain will be evaluated using a numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain, and 10 points representing the sharpest pain.
Incidence of lidocaine toxicity within 72 hours after surgery | within 72 hours after surgery
  the occurrence of one or more adverse events including tingling/pins and needles, especially around the eyes and mouth, ringing in the ears, dizziness, visual disturbances, and metallic taste.
Quality of Recovery Scale Score (QoR-15) at 24, 48, and 72 hours after surgery | 24, 48, and 72 hours after surgery
  The global QoR-15 score ranges from 0 to 150 and is categorized as five quality of recovery dimensions, including physical comfort (5 items), emotional state (4 items), psychological support (2 items), physical independence (2 items), and pain (2 items). Each piece is graded using an 11-point Likert scale. The QoR is classified according to the QoR-15 score as excellent (QoR-15 > 135), good (122 ≤ QoR-15 ≤ 135), moderate (90 ≤ QoR-15 ≤ 121) and poor (QoR-15 < 90).
Bowel function recovery | From the end of surgery to discharge, up to 1 week
  defined as the time to first defecation or the time to first flatus
Incidence of adverse reactions to opioids within three days after surgery | within three days after surgery
  It is defined as if patients happened any constipation, nausea, vomiting, drowsiness, dizziness, itchy skin, confusion, respiratory depression, etc.
The incidence of a composite of postoperative pulmonary complications during hospitalization | from the end of surgery to discharge, up to 1 week
  defined as positive if any component developed before discharge after surgery; These complications included respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, or aspiration pneumonitis
Length of hospital stay | from the end of surgery to discharge, up to 1 month.
  determined by the number of days from admittance to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Chunling, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No